CLINICAL TRIAL: NCT05457738
Title: Home-based Exercice Therapy for Patients With Intermittent Claudication Using a New Smartphone Application : a Monocentric Randomized Study
Brief Title: Home-based Exercice Therapy for Patients With Intermittent Claudication Using a New Smartphone Application
Acronym: APAISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PA22075
Record Dates: First submitted 2022-06-30; First posted 2022-07-14 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Intermittent Claudication
Keywords: Intermittent claudication; peripheral arterial disease; supervised exercise therapy; home-based exercise; smartphone medical application
MeSH Terms: conditions — Intermittent Claudication; Peripheral Arterial Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients randomized to using the smartphone app (Experimental)
  Interventions: Other: E-REVA® app
- patients randomized to not using the smartphone app (Active Comparator)
  Interventions: Other: No E-REVA® app

INTERVENTIONS:
Other: E-REVA® app — Use of a smartphone app designed for home-based exercise therapy of patients with intermittent claudication. App's name is E-REVA®.
  Arms: patients randomized to using the smartphone app
Other: No E-REVA® app — No use smartphone
  Arms: patients randomized to not using the smartphone app

SUMMARY:
The main characteristic of PAD is to limit physical activity by the appearance of claudication of the lower limbs which limits the walking distance, or the maximum distance traveled by the patient before the pain forces to stop. In daily practice, the walking distance is rarely measured at the time of treatment.

Walking rehabilitation is the first-line treatment for these patients (class 1 recommendation from the AHA 2005 and the ESC 2017 with level A evidence). According to the recommendation, a walking session must last at least 30 minutes at the rate of 3 sessions per week for a minimum of 6 months.

Walking rehabilitation should be systematically offered to all claudicating patients, whether operated on or not. It is often sufficient for mild claudication with a walking distance of more than 500 meters. Surgery should be reserved for patients in whom rehabilitation has failed and in whom the claudication is severe (walking distance less than 500 meters). Surgical intervention should not replace rehabilitation, but should be complementary.

Supervised rehabilitation in specialized centers is rarely offered because it is not easily available and involves additional expenses and constraints for the patient (transport, fewer work periods for active patients, etc.). In the absence of specialized center, simple advice is most often given to the patient, who then only has to rely on his personal motivation: this is the so-called "go home and walk".

Therefore, access to well-conducted rehabilitation is a fundamental element of the management of patients with intermittent claudication, which is currently lacking. In the age of digital health, it is necessary to develop innovative tools allowing self-rehabilitation of the patient in addition with remote monitoring by the doctor.

Recent studies have validated and highlighted the interest of using GPS technology for the evaluation of walking activity in claudicants. To date, there are 2 published examples of smartphone applications developed specifically for exercise rehabilitation. The main shortcomings of the solutions proposed in these publications are:

* The need to buy a specific GPS box
* Discomfort for the patient to carry the box either in a backpack or over the shoulder
* The lack of means for the patient to indicate the precise moment when the pain appears
* And consequently the absence of clinical analysis centered on the symptom "walk induced pain" Consumer smartphone applications for GPS activity tracking are not intended for medical use and do not indicate when pain occurs.

In this study, the University Hospital of REIMS will establish a scientific collaboration with the company VascInnove® for the use of a smartphone application, called E-REVA® which offers:

* an assessment of walking activity and claudication parameters (appearance of pain, walking distance, recovery time after pain, total distance travelled, walking speed, etc.)
* help with self-rehabilitation
* quality of life and walking questionnaires

The main innovation is the presence of a button allowing the patient to indicate when the pain appears. The patient will be able to have access via the smartphone application to his statistics and the evolution of his performance over time. The prescribing practitioner will have access, via a secure website, to the statistics of his patient, to whom he will be able to give personalized advice during follow-up consultations.

The aim of this study is to carry out a single-centre prospective randomized stratified study (depending on whether or not patient has been revascularized) in patients with intermittent claudication who will or will not use the rehabilitation assistance smartphone application, seen in consultation for vascular surgery and vascular medicine at the University Hospital of Reims.

ELIGIBILITY:
inclusion criteria :

* - Patient over 18 years old
* Patient with claudication on PAD for more than 3 months
* IPS (systolic pressure index) less than 0.90 at the level of the diseased limb
* Absence of pathology limiting walk other than PAD
* Patient having benefited from an arterial ultrasound of the lower limbs demonstrating arterial lesion
* Absence of myocardial infarction over the last 6 months
* Absence of cardiac pathology requiring surgery
* Absence of angina
* Patient affiliated or entitled to a social security system
* Patient having given his free and written consent

exclusion criteria :

* Patient who has not benefited from an arterial ultrasound of the lower limbs
* All contraindications to treadmill events:

  * Myocardial infarction within the last 6 months
  * angina
  * Symptomatic tight aortic valve stenosis
  * Pathology limiting walk other than PAD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2028-05-19 (Estimated); Study Completion 2028-05-19 (Estimated)

PRIMARY OUTCOMES:
maximal walking distance on treadmill test | 3 months
maximal walking distance on treadmill test | 12 months

SECONDARY OUTCOMES:
Quality of life assessment VascuQol-6 | 6 months
Walking Impairment Questionnaire | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France